CLINICAL TRIAL: NCT06358664
Title: The Effect of Caffeine Consumption on Cataract Formation After Pars Plana Vitrectomy: a Comparative Study
Brief Title: Caffeine and Cataract After Pars Plana Vitrectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Principal Investigator, Vienna Institute for Research in Ocular Surgery
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Caffeine Vitrectomy
Record Dates: First submitted 2024-04-04; First posted 2024-04-10 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Cataract
Keywords: Pars plana vitrectomy; Caffeine; Retinal detachment; Macular Pucker
MeSH Terms: conditions — Cataract; Retinal Detachment; Epiretinal Membrane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caffeine consumption (Experimental): Patients with regular caffeine consumption needing pars plana vitrectomy
  Interventions: Procedure: Pars plana vitrectomy
- No caffeine consumption (Experimental): Patients with regular caffeine consumption needing pars plana vitrectomy
  Interventions: Procedure: Pars plana vitrectomy

INTERVENTIONS:
Procedure: Pars plana vitrectomy — Standard pars plana vitrectomy will be performed

SUMMARY:
Assessment of cataract development in patients with regular caffeine consumption and those without caffeine consumption after pars plana vitrectomy.

DETAILED DESCRIPTION:
Vitrectomy is a frequently used surgical procedure in ophthalmology for various indications like retinal detachment repair or macular pucker peeling. Amongst others, accelerated cataract development in phakic patients is a known complication after vitrectomy. A previous study found that especially patients receiving gas tamponade are at increased risk for postoperative cataract development. The assumed mechanism behind this finding is that vitrectomy leads to an increased partial pressure of O2 in the human vitreous - similar to that observed in posterior vitreous detachment - subsequently leading to accelerated lens opacification. Therefore, a possible target of cataract prevention is the inhibition of oxygen radical formation. One known antioxidant agent inhibiting oxygen radical formation is caffeine. For instance, in-vitro studies showed that caffeine consumption can reduce cataract development in ultraviolet (UV)-radiation-exposed rats and human lens epithelial cells through its capability of inhibiting oxygen radical formation. These in-vitro studies support the findings of epidemiological studies that caffeine also in-vivo has the potential to reduce cataractogenesis. Conflating the previous findings of accelerated cataract formation after vitrectomy and the preventive properties of caffeine for cataract development, there may be a benefit for patients regularly consuming caffeine-containing beverages like coffee undergoing vitrectomy regarding postoperative cataract formation.

Therefore, the aim of this comparative study is to investigate if patients undergoing small gauge pars plana vitrectomy regularly consuming caffeine have lower postoperative significant cataract formation rates than patients not consuming caffeine.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Written informed consent
* No previous cataract surgery in the study eye
* Scheduled small gauge vitrectomy with intraoperative gas tamponade (SF6 or C3F8) due to retinal detachment or macular hole repair
* No regular caffeine consumption (drinking not more than one cup of a caffeine- containing beverage [e.g. coffee, energy drinks] at a maximum of two days per week during the past year)

Exclusion Criteria:

* Intake of systemic or topical corticosteroids within 3 months before study screening
* Increased risk for postoperative cataract development, for example due to ocular trauma in the history
* Severe cataract (LOCS III grading of any cataract form >2) in the study eye at pre- study screening
* Scheduled phacovitrectomy in the study eye
* Participation in any clinical trial three month before study screening
* Ocular surgeries six month before study screening

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Significant cataract formation at year 1 | 12 months
  Frequency of significant cataract formation one year after vitrectomy in study eyes as compared to control eyes

SECONDARY OUTCOMES:
Significant cataract formation at month 6 | 12 months
  Frequency of significant cataract formation 6 months after vitrectomy in study eyes as compared to control eyes
Distance corrected visual acuity (DCVA) | 12 months
  DCVA at all study visits in study eyes as compared to control eyes

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, Prim. Dr., Principal Investigator — Vienna Institute for Research in Ocular Surgery (VIROS), Hanusch Krankenhaus
Locations (1):
- Vienna Institute for Research in Ocular Surgery (VIROS), Hanusch Hospital, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No